CLINICAL TRIAL: NCT02935218
Title: Parenting Skills for Mothers With Borderline Personality Disorder: A Newly Developed Group Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Dr. Charlotte Rosenbach, Dr, Freie Universität Berlin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RenRos01
Record Dates: First submitted 2016-08-30; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-09

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parenting Skills for Mothers with BPD (Other): single-arm study
  Interventions: Behavioral: Parenting Skills for Mothers with BPD

INTERVENTIONS:
Behavioral: Parenting Skills for Mothers with BPD — The cognitive-behavioral Group Training for mothers with BPD consists of 12 weekly sessions promoting parenting skills including primary needs of children, stress and stress management, dealing with conflicts, mindfulness, emotion regulation, routine and flexibility, the role of the body in parenting, basic assumptions about parenting, and self-care.

SUMMARY:
N=15 mothers with Borderline Personality Disorder who had young children (aged 0-6 years) participated in a 12-week training program. To estimate the participants' impairment, parental stress and psychological distress were assessed before the training. After the training, participants and trainers were asked to provide feedback regarding the valuation of and the changes due to the training.

ELIGIBILITY:
Inclusion Criteria:

* Borderline diagnosis in mothers
* Infants between 6 months and 6 years
* Mothers and their children must be in regular contact with each other

Exclusion Criteria:

* Acute child endangerment
* Maternal acute suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
written feedback | 12 weeks
  the participants provide written feedback regarding the changes due to the parental skills training

IPD SHARING:
Plan to Share IPD: No
qualitative data not suitable for sharing

REFERENCES:
- [Derived] Renneberg B, Rosenbach C. "There is not much help for mothers like me": Parenting Skills for Mothers with Borderline Personality Disorder - a newly developed group training program. Borderline Personal Disord Emot Dysregul. 2016 Dec 1;3:16. doi: 10.1186/s40479-016-0050-4. eCollection 2016. PMID 27980787